CLINICAL TRIAL: NCT04782869
Title: Personalized Multichannel Transcranial Direct Current Electrical Stimulation (tDCS) in Drug-resistant Epilepsy: Evaluation of Therapeutic and Neurophysiological Effects
Brief Title: Transcranial Direct Current Electrical Stimulation (tDCS) in Drug-resistant Epilepsy
Acronym: GALVANI PS-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-55; ID-RCB (Other: 2020-A02861-38)
Record Dates: First submitted 2021-02-26; First posted 2021-03-04 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Epilepsy
Keywords: pharmaco-resistant epilepsy; transcranial stimulation; SEEG
MeSH Terms: conditions — Epilepsy | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS (transcranial direct current stimulation) (Experimental): Patient will be treated for 3 cycles. A cycle is composed of 5 bi-sessions (one per day) of 20 minutes each.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — Patients will be treated using Starstim 8 device, a device allowing to perform transcranial direct current stimulation. The position of electrodes will be personalized based on the localization of the epileptogenic zone.

SUMMARY:
This project aims to conduct a pilot study based on the targeting of the epileptogenic zone previously localized very precisely by stereoelectroencephalography (SEEG). SEEG is used as part of the pre-surgical assessment. It consists, thanks to the intracerebral implantation of electrodes in the brain of patients, to perform an intracerebral electrophysiological recording and thus to precisely explore the epileptogenic regions.

In order to study the neuromodulatory and therapeutic effects of tDCS on epileptic brains, non-invasive techniques for measuring electrophysiological brain activity such as magnetoencephalography (MEG) and high-resolution electroencephalography (HR EEG) will be used.

Finally, since epilepsy is considered to be a disorder of brain functional networks associated with disturbed brain connectivity, the effects of tDCS on cortical excitability by studying the variations in functional connectivity induced by stimulation will be studied.

ELIGIBILITY:
Inclusion Criteria:

* - Age: Older than 12 years old
* Patients with drug-resistant focal epilepsy with no surgical indication or with a previous surgical failure or refusing surgery.
* SEEG previously performed before inclusion with an adequate definition of the epileptogenic zone
* A clinical or research MRI scan that is suitable for navigated brain stimulation (NBS) and definition of target area.
* Number of seizures >3/month during the baseline (before the first session of tDCS treatment), for at least 3 months
* Have stable medications for the whole study duration and few weeks before
* Total IQ>65
* Be able to understand, speak and write in French
* Patient, parents or legally representative who have given written informed consent to allow the study data collection procedures,
* Be a beneficiary of affiliated to a health insurance plan

Exclusion Criteria:

* - Generalized epilepsy
* Presenting contraindication to MRI, a serious intercurrent pathology, a progressive brain tumor
* Skin conditions (e.g., eczema, lesion)
* Any cranial metal implants (excluding <1 mm thick epicranial titanium skull plates and dental fillings) or medical devices (i.e. cardiac pacemaker, deep brain stimulator, medication infusion pump, cochlear implant).
* Previous surgeries opening the skull leaving skull defects capable of allowing the insertion of a cylinder with a radius greater or equal to 5 mm.
* Metal inside the head (outside the mouth) such as shrapnel, surgical clips
* Patient currently participating in another clinical trial or having participated in a clinical trial in the month prior to inclusion.
* Any condition that makes the study subject, in the opinion of the investigator, unsuitable for the study.
* Person protected by articles L1121-5, L1121-6 and L1121-8 of Public Health Code (pregnant or breastfeeding woman, deprived of liberty by judicial decision, situations of social fragility, adults unable or unable to express their consent).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Seizure frequency | Comparison between baseline and month 2
  Percentage of change of seizures frequency
Seizure frequency | Comparison between baseline and month 4
  Percentage of change of seizures frequency
Seizure frequency | Comparison between baseline and month 6
  Percentage of change of seizures frequency
Seizure frequency | Comparison between baseline and month 8
  Percentage of change of seizures frequency

SECONDARY OUTCOMES:
Depression | Comparison between baseline and month 8
  Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) - score to 6 to 24, higher values mean worse outcome
Anxiety disorders | Comparison between baseline and month 8
  Generalized Anxiety Disorder-7 (GAD-7) - score between 0 to 21, higher values mean worse outcome
Seizures evaluation | Comparison between baseline and month 8
  National Hospital Seizure Severity Scale (NHS3) - score 1 to 31, higher values mean worse outcome
Brain functional connectivity | Comparison between day 1 and day 5 of each session
  National Hospital Seizure Severity Scale (NHS3) score 1 to 31, higher values mean worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier Arnaud, Study Director — AP-HM
Locations (1):
- Service d'Epileptologie et de Rythmologie Cérébrale, Marseille, France

IPD SHARING:
Plan to Share IPD: No